CLINICAL TRIAL: NCT07184047
Title: Effectiveness of G8 and VES-13 Frailty Scales in Predicting Chemotherapy Toxicity in Older Patients With Gastrointestinal Cancers: A Prospective Observational Study
Brief Title: Frailty Scales for Predicting Chemotherapy Toxicity in Older Adults With Gastrointestinal Cancers
Acronym: TOX-FRAIL
Status: Active, not recruiting | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Galip Can Uyar, Medical Oncologist Specialist, Ankara Etlik City Hospital
Other Study IDs: AEŞH-BADEK-2024-039; AEŞH-BADEK-2024-039 (Other: Ankara Etlik City Hospital Scientific Research Ethics Committee)
Record Dates: First submitted 2025-09-14; First posted 2025-09-19 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Cancers; Frailty; Sarcopenia in Elderly; Malnutrition Elderly; Toxicity Due to Chemotherapy; Colorectal Cancer; Gastric Cancer (GC); Pancreatic Cancer Resectable; Biliary Tract Cancer; Esophageal Cancer (EsC); Older Adults (65 Years and Older)
Keywords: Frailty; G8 Screening Tool; VES-13; Chemotherapy Toxicity; Older adults; sarcopenia; malnutrition; Nutritional Assessment (MNA-SF); Activities of Daily Living (ADL, IADL); ECOG Performance Status; Supportive Oncology; Geriatric Oncology
MeSH Terms: conditions — Gastrointestinal Neoplasms; Frailty; Colorectal Neoplasms; Stomach Neoplasms; Biliary Tract Neoplasms; Esophageal Neoplasms; Sarcopenia; Malnutrition; Sarcoglycanopathies | interventions — Chemotherapy, Adjuvant; Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adjuvant Chemotherapy Cohort: Older patients (≥65 years) with non-metastatic or locally advanced gastrointestinal cancers receiving standard adjuvant chemotherapy (e.g., FOLFOX, CAPEOX, FOLFIRI, FOLFOXIRI, FOLFIRINOX, capecitabine, gemcitabine, 5-FU/leucovorin, or oxaliplatin-based regimens). Patients will undergo frailty, nutritional, sarcopenia, functional, and performance status assessments at baseline, 3 months, and at the end of chemotherapy. Treatment will follow routine clinical practice, and no investigational intervention will be administered.
  Interventions: Other: Adjuvant Chemotherapy (Standard of Care)

INTERVENTIONS:
Other: Adjuvant Chemotherapy (Standard of Care) — Patients aged 65 years and older with non-metastatic or locally advanced gastrointestinal cancers will receive standard adjuvant chemotherapy regimens as part of routine clinical practice. Regimens may include FOLFOX, CAPEOX, FOLFIRI, FOLFOXIRI, FOLFIRINOX, capecitabine, gemcitabine, 5-FU/leucovorin, or oxaliplatin-based combinations, depending on tumor type and physician decision.
  No investigational drugs or experimental interventions are administered. The study is observational, and all treatments follow standard of care.

SUMMARY:
This study evaluates the effectiveness of the G8 and VES-13 frailty scales in predicting chemotherapy-related toxicity in older patients with gastrointestinal cancers receiving adjuvant chemotherapy. Older adults are more vulnerable to treatment-related side effects due to age-related declines in physiological reserve. Early identification of frailty may help individualize treatment decisions and optimize supportive care.

This is a prospective, single-center, observational study conducted at Ankara Etlik City Hospital. A total of 72 patients aged 65 years and older with non-metastatic or locally advanced gastrointestinal cancers scheduled for adjuvant chemotherapy will be included.

Frailty, sarcopenia, nutritional status, functional independence, and performance status will be assessed at baseline, 3 months, and at the end of chemotherapy.

The primary aim is to determine the predictive value of G8 and VES-13 scores for chemotherapy-related toxicity. Secondary aims include exploring the associations between frailty, nutritional status, sarcopenia, daily living activities, and treatment tolerance. Additionally, one-year progression-free survival (PFS) and overall survival (OS) will be analyzed.

DETAILED DESCRIPTION:
Background

Gastrointestinal (GI) cancers in older adults are often accompanied by frailty, malnutrition, and functional decline, which increase the risk of chemotherapy-related toxicity. While chemotherapy in the adjuvant setting is standard of care, toxicities may impair quality of life and adherence in this vulnerable population. Validated frailty screening tools may improve risk stratification and supportive care strategies.

Study Design

Type: Prospective, observational, single-center, non-randomized study

Site: Ankara Etlik City Hospital, Department of Medical Oncology

Target enrollment: 72 patients

Population: Patients ≥65 years with non-metastatic or locally advanced GI cancers (esophageal, gastric, colorectal, pancreatic, or biliary tract) scheduled for adjuvant chemotherapy only

Exclusion: ECOG PS ≥3, severe frailty at baseline, patients planned for chemoradiotherapy, or those receiving neoadjuvant chemotherapy

Timeline:

First patient in: January 15, 2024

Accrual closure: January 1, 2025

Final data collection (PFS/OS): January 1, 2026

Assessments

Patients will be assessed at baseline, mid-treatment (~3 months), and at the end of chemotherapy (~6 months). All instruments have been validated in Turkish populations:

G8 Screening Tool

Range: 0-17

Cut-off ≤14 = frailty risk

VES-13 (Vulnerable Elders Survey-13)

Range: 0-13

Cut-off ≥3 = frailty

SARC-F (Sarcopenia screening tool)

Range: 0-10

Cut-off ≥4 = probable sarcopenia

Mini Nutritional Assessment - Short Form (MNA-SF)

12-14 = normal nutrition

8-11 = at risk

0-7 = malnutrition

Katz Index of Activities of Daily Living (ADL)

Range: 0-6 (higher = more independence)

Lawton-Brody Instrumental Activities of Daily Living (IADL)

Range: 0-8 (higher = more independence)

ECOG Performance Status

Range: 0-5 (higher = worse functional state)

Outcomes

Primary outcome:

Predictive value of G8 and VES-13 for grade ≥2 chemotherapy-related toxicity (CTCAE v5.0)

Secondary outcomes:

Associations between frailty and sarcopenia, nutrition, functional independence, and ECOG

One-year Progression-Free Survival (PFS)

One-year Overall Survival (OS)

Statistical Analysis

Categorical variables will be analyzed using Chi-square or Fisher's exact test. Continuous variables will be compared using t-test or Mann-Whitney U test, depending on distribution. Survival analyses (PFS, OS) will be estimated with Kaplan-Meier method. A p-value <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Histologically confirmed non-metastatic or locally advanced gastrointestinal cancers (esophageal, gastric, colorectal, pancreatic, biliary tract)
* Planned to receive adjuvant chemotherapy (standard regimens such as FOLFOX, CAPEOX, FOLFIRI, FOLFOXIRI, FOLFIRINOX, capecitabine, gemcitabine, 5-FU/leucovorin, or oxaliplatin-based regimens)
* ECOG Performance Status 0-2
* Ability to complete frailty and functional assessment questionnaires (G8, VES-13, SARC-F, MNA-SF, Katz ADL, Lawton-Brody IADL)
* Signed informed consent

Exclusion Criteria:

* ECOG Performance Status ≥3
* Patients planned for neoadjuvant chemotherapy or chemoradiotherapy
* Prior systemic chemotherapy or radiotherapy for the same cancer diagnosis
* Severe cognitive impairment preventing questionnaire completion
* Patients with advanced frailty at baseline screening
* Concurrent enrollment in another interventional clinical trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of at least 72 older patients (≥65 years) with non-metastatic or locally advanced gastrointestinal cancers who are scheduled to receive standard adjuvant chemotherapy at Ankara Etlik City Hospital, Department of Medical Oncology. Patients will be assessed for frailty, sarcopenia, nutritional status, functional independence, and performance status at baseline, 3 months, and 6 months during chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of the Geriatric-8 (G8) and the Vulnerable Elders Survey-13 (VES-13) Frailty Scales for Chemotherapy-Related Toxicity | Baseline, 3 months after chemotherapy initiation, and 6 months (end of adjuvant chemotherapy)
  The predictive ability of the G8 (score 0-17; cut-off ≤14) and VES-13 (score 0-13; cut-off ≥3) frailty screening tools in identifying older patients (≥65 years) with gastrointestinal cancers who are at risk of developing grade ≥2 chemotherapy-related toxicity. Toxicities will be assessed according to CTCAE version 5.0 and reported as the proportion (%) of patients with grade ≥2 events. Both frailty tools have validated Turkish versions.

SECONDARY OUTCOMES:
Correlation of Frailty Scores with the Strength, Assistance with walking, Rise from a chair, Climb stairs, and Falls (SARC-F) Questionnaire | Baseline, 3 months after chemotherapy initiation, and 6 months (end of adjuvant chemotherapy)
  Correlation of Geriatric-8 and Vulnerable Elders Survey-13 frailty scores with sarcopenia risk assessed by the Strength, Assistance with walking, Rise from a chair, climb stairs, and Falls (SARC-F) questionnaire (range 0-10; cut-off ≥4; validated in Turkish). Scores will be reported as points on the scale.
Correlation of Frailty Scores with the Mini Nutritional Assessment - Short Form (MNA-SF) Questionnaire | Baseline, 3 months after chemotherapy initiation, and 6 months (end of adjuvant chemotherapy)
  Correlation of Geriatric-8 and Vulnerable Elders Survey-13 frailty scores with nutritional risk assessed by the Mini Nutritional Assessment - Short Form (MNA-SF) questionnaire (range 0-14; categories: 12-14 = normal, 8-11 = risk, 0-7 = malnutrition; validated in Turkish). Scores will be reported as points on the scale.
Correlation of Frailty Scores with the Katz Index of Activities of Daily Living (ADL) | Baseline, 3 months after chemotherapy initiation, and 6 months (end of adjuvant chemotherapy)
  Correlation of Geriatric-8 and Vulnerable Elders Survey-13 frailty scores with functional independence assessed by the Katz Index of Activities of Daily Living (ADL; range 0-6; validated in Turkish). Scores will be reported as points on the scale.
Correlation of Frailty Scores with the Lawton-Brody Instrumental Activities of Daily Living (IADL) Scale | Baseline, 3 months after chemotherapy initiation, and 6 months (end of adjuvant chemotherapy)
  Correlation of Geriatric-8 and Vulnerable Elders Survey-13 frailty scores with functional independence assessed by the Lawton-Brody Instrumental Activities of Daily Living (IADL) scale (range 0-8; validated in Turkish). Scores will be reported as points on the scale.
Correlation of Frailty Scores with the Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline, 3 months after chemotherapy initiation, and 6 months (end of adjuvant chemotherapy).
  Correlation of Geriatric-8 and Vulnerable Elders Survey-13 frailty scores with the Eastern Cooperative Oncology Group (ECOG) Performance Status (range 0-5; validated in Turkish). Scores will be reported as points on the scale.
Overall Survival (OS) | 12 months after chemotherapy initiation
  Overall survival will be defined as the time from chemotherapy initiation to death from any cause, measured in months.
Progression-Free Survival (PFS) | 12 months after chemotherapy initiation.
  Progression-free survival will be defined as the time from chemotherapy initiation to disease progression or death from any cause, measured in months.

CONTACTS AND LOCATIONS:
Overall Officials: Galip Can Uyar, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Medical Oncology Department, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No